CLINICAL TRIAL: NCT05262868
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Affective Symptoms in Patients Suffering From Dementia: a Randomised Clinical Trial
Brief Title: rTMS for the Treatment of Affective Symptoms in Patients Suffering From Dementia
Acronym: rTMS-PSYGER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof Armin von Gunten, Professor, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-D0067
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Magnetic stimulus intensity of 80% of the motor threshold applied at the frequency of 20 Hz over the left DLPFC with a total number of pulses of 1200 / treatment session for a total of 5 sessions /week for 3 consecutive weeks
  Interventions: Device: rTMS
- Sham (Placebo Comparator): Sham procedure implies the use of a "sham" coil of exactly the same dimension and appearance as the one used for the effective treatment. This sham coil is made for research purposes by the producing company and used in accordance with the instructions for use, which explicitly mention it (cf. instruction manual page 34: Stimulation Coil DuoMAG 70BFP (70BFP1, 70BFP2), typical use for blinded studies).
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — The stimulus intensity will be 80% of the motor threshold and the frequency will be 20 Hz for all patients. The total number of pulses will be 1200 for a single treatment session. We plan a total of 15 sessions distributed over 5 days a week for 3 consecutive weeks.

SUMMARY:
This is a monocentric prospective, randomized, double-blind placebo-controlled study. It is designed to evaluate the superiority of the rTMS over sham treatment of depressive symptoms in the context of dementia. It is aimed at a population ≥ 65 years old, with affective BPSD. We wish to recruit 44 participants, with an estimated rate of potential drop out of 20%. Patients will be randomly assigned to the sham or rTMS group. The sham stimulation reproduces the procedure in all the steps, has the same duration and differs exclusively by the device setting. After inclusion, both groups will receive 15 sessions distributed over 5 days a week for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by their and their proxy's signature (Appendix Informed Consent Form)
* Consent for MRI
* Age ≥ 65 years
* Clinical dementia Rating Scale (CDR) ≥ 1
* NPI-Q Σ (*Anxiety + * Apathy/Indifference + * Dysphoria/Depression) ≥ 3
* Cornell Scale for Depression in Dementia (CSDD) ≥ 10

Exclusion Criteria:

* History of schizophrenia, bipolar disorder, schizoaffective disorder
* History of macroscopic stroke.
* Unstable somatic pathologies
* Insufficient collaboration for the rTMS procedure
* Drug freeness or drug adjustment as clinically required is not an exclusion criterion.
* The proxy refuses to give consent in case of lack of capacity, or in any case where the participant expresses a wish not to participate/continue in the study.
* Any contraindications to performing an MRI (cf CRF) and rTMS (aneurysm clips or coils, stents in the neck or brain, deep brain stimulators, electrodes to monitor brain activity, metal implants in the ears and eyes, facial tattoos with metallic or magnetically sensitive ink) procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Cornell Scale for Depression in Dementia (CSDD) | from baseline to day 20
  Mood assessment tool

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | from baseline to day 20
  Cognitive assessment tool
NPI-Q | from baseline to day 20
  Behavioural assessment tool for demented patients
The ratio of patients who completed the study and drop-outs due to non-compliance | During all the study period
  Compliance assessment tool
Possible changes of structural MRI before as compared to after the treatment | from baseline to day 20
  quantitative structural MRI protocol allowing for an optimal segmentation - resolution of grey versus white matter including cortical and sub-cortical brain structures.

CONTACTS AND LOCATIONS:
Overall Officials: Armin von Gunten, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Supaa - Chuv, Prilly, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No